CLINICAL TRIAL: NCT01275521
Title: Study of the Effectiveness and the Tolerance of Intraprostatic A-botulinic Toxin Injection, in the Treatment of Symptomatic Benign Prostate Hypertrophy.
Brief Title: A-botulinic Toxin for Symptomatic Benign Prostate Hypertrophy
Acronym: PROTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2010/39
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BONT-A intra-prostatic injection (Experimental)
  Interventions: Drug: BONT-A intra-prostatic injection
- optimized medical BPH treatment (Active Comparator)
  Interventions: Drug: Optimized medical BPH treatment

INTERVENTIONS:
Drug: BONT-A intra-prostatic injection — • Intra prostatic injection of 200 IU of BONT-A (2 x 100 IU to dilute in 10 cc salted serum), divided into 4 injections, 2 in each prostate lobe for a volume intra injected 2.5 cc per site.
  Interruption of the medical therapy 1 month after the injection;
  Arms: BONT-A intra-prostatic injection
Drug: Optimized medical BPH treatment — Optimization of the medical therapy according to recent guidelines
  Arms: optimized medical BPH treatment

SUMMARY:
BPH is very common in elderly men, it is a stromal as well as epithelial invasion of the prostatic gland. Due to an imbalance between growth and apoptosis cellular mechanisms that are not fully elucidated. It is the same for symptomatology and urodynamic obstruction without clear identification of the part which is due to static phenomena (volume increase) and dynamic reports (α 1-receptor action). That explains the multiplicity of treatments and the difficulty of therapeutic indications between monitoring, medical treatment, and surgical operation. Experimental studies of BONT-A intra prostatic injection on animal and human models, have shown efficacy in BPH cell apoptosis, decrease in cell growth and decline in the number of adrenergic α1 receptors.

Many studies in humans show therapeutic efficacy leading to a possible use of BONT-A as mini invasive treatment of symptomatic BPH, as an alternative to medical or surgical treatment.

PROTOX study proposes to evaluate tolerance and effectiveness of the intra-prostatique BONT-A injection in the treatment of symptomatic BPH.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 50 to 85;
* Obstructive or irritative urinary symptomatology linked to a BPH;
* Score IPSS moderate to severe (8-19: moderate; 20-35: severe) or IPSS ≤ 7 in patient medically treated for symptomatic BPH;
* Increase in prostate volume on the rectal touch or ultrasound;
* Free consent, informed and written, dated and signed by the patient and the investigator (at the latest the day inclusion and before any examination requires the study);
* Subject affiliate or beneficiary of a social protection

Exclusion Criteria:

* stenosis of the urethra confirmed by endoscopic or radiological examination;
* prostate cancer suspicion;
* medical past history of surgery, radiotherapy or pelvic trauma (, breach of the urethra, pubic symphysis disjunction);
* surgical resection of the prostate (adenomecty);
* clinical or paraclinical signs of vesical sphincterial disynergia; chronic urinary retention > 500 ml;
* BPH complications making surgery necessary: effects on the upper urinary tract: dilatation or renal obstructive insufficiency, bladder stones or diverticula.
* patient previously treated by botulic toxin (whatever injection site);
* Persons unable to understand the course of the study.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2015-04-28 (Actual); Study Completion 2015-04-28 (Actual)

PRIMARY OUTCOMES:
Evaluation of the patient with auto-questionnaire IPSS urinary symptomatology: questions 1 to 7 (0 to 35 score). | 4 months

SECONDARY OUTCOMES:
IPSS question 8 (score 0 to 6) | 18 months
Uroflowmetry (Qmax in ml/s) | 18 months
• measure the post-voiding residue assessed by supra pubic ultrasound or urinary drainage | 18 months
measure of prostate volume assessed by endo-rectal ultrasound | 18 months
measurement of the erectile function by auto questionnaire IIEF-5 (0 to 24 score) | 18 months
urinary continence Evaluation by ICS 1 (0 to 23 score) and ICS 2 (0 to 12 score) | 18 months
bladder emptying mode (spontaneous or permanent probe) | 18 months
specific treatment for BPH (alpha blocking, 5 alpha reductase inhibitor and/or phytotherapy) | 18 months
Urinary retention | 18 months
Surgical treatment | 18 months
profile of gene and protein expression on the first urine flow after prostate massage | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire ROBERT, MD, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, MD, Study Chair — University Hospital, Bordeaux
Locations (11):
- France (11):
  - Service d'Urologie - CH du Pays d'Aix - Avenue de Tamaris, Aix-en-Provence
  - Service d'Urologie, CHU d'Angers 4, rue Larrey, Angers
  - Service d'urologie, Groupe Hospitalier Pellegrin, place Amélie Raba Léon, Bordeaux
  - Service d'urologie - APHP Henri Mondor - 51, avenue du Maréchal de Lattre de Tassigny, Créteil
  - Service d'urologie - CHU de Limoges - 2, avenue Martin Luther King, Limoges
  - Service d'urologie - Hôpital de la Conception - 147 boulevard Baille, Marseille
  - Clinique Mutualiste Beausoleil, Montpellier
  - Service d'Urologie - APHP Hopital Cochin - 27, Rue du faubourg Saint Jacques, Paris
  - Service d'Urologie - APHP Hôpital Saint Louis - 1, avenue Claude-vellefaux, Paris
  - Service d'Urologie - Hospices Civls de Lyon - 165 chemin du grand Revoyet, Pierre-Bénite
  - Service d'urologie - CHRU Strasbourg - BP 426, Strasbourg

REFERENCES:
- [Background] Costa P, Ben Naoum K, Boukaram M, Wagner L, Louis JF. [Benign prostatic hyperplasia (BPH): prevalence in general practice and practical approach of French general practitioners. Results of a study based on 17,953 patients]. Prog Urol. 2004 Feb;14(1):33-9. French. PMID 15098749
- [Background] Rhodes PR, Krogh RH, Bruskewitz RC. Impact of drug therapy on benign prostatic hyperplasia-specific quality of life. Urology. 1999 Jun;53(6):1090-8. doi: 10.1016/s0090-4295(99)00041-2. PMID 10367833
- [Background] Isaacs JT, Coffey DS. Etiology and disease process of benign prostatic hyperplasia. Prostate Suppl. 1989;2:33-50. doi: 10.1002/pros.2990150506. PMID 2482772
- [Background] Chute CG, Stephenson WP, Guess HA, Lieber M. Benign prostatic hyperplasia: a population-based study. Eur Urol. 1991;20 Suppl 1:11-7. doi: 10.1159/000471739. PMID 1722154
- [Background] McConnell JD. The pathophysiology of benign prostatic hyperplasia. J Androl. 1991 Nov-Dec;12(6):356-63. PMID 1722791
- [Background] Barrack ER, Bujnovszky P, Walsh PC. Subcellular distribution of androgen receptors in human normal, benign hyperplastic, and malignant prostatic tissues: characterization of nuclear salt-resistant receptors. Cancer Res. 1983 Mar;43(3):1107-16. PMID 6186370
- [Background] Marcelli M, Shao TC, Li X, Yin H, Marani M, Denner L, Teng B, Cunningham GR. Induction of apoptosis in BPH stromal cells by adenoviral-mediated overexpression of caspase-7. J Urol. 2000 Aug;164(2):518-25. PMID 10893637
- [Background] Colombel M, Vacherot F, Diez SG, Fontaine E, Buttyan R, Chopin D. Zonal variation of apoptosis and proliferation in the normal prostate and in benign prostatic hyperplasia. Br J Urol. 1998 Sep;82(3):380-5. doi: 10.1046/j.1464-410x.1998.00752.x. PMID 9772874
- [Background] Radlmaier A, Eickenberg HU, Fletcher MS, Fourcade RO, Reis Santos JM, van Aubel OG, Bono AV. Estrogen reduction by aromatase inhibition for benign prostatic hyperplasia: results of a double-blind, placebo-controlled, randomized clinical trial using two doses of the aromatase-inhibitor atamestane. Atamestane Study Group. Prostate. 1996 Oct;29(4):199-208. doi: 10.1002/(SICI)1097-0045(199610)29:43.0.CO;2-7. PMID 8876703
- [Background] Frick J. [Pathophysiology of benign prostatic hyperplasia]. Wien Med Wochenschr. 1996;146(8):158-60. German. PMID 8767399
- [Background] Hieble JP, Boyce AJ, Caine M. Comparison of the alpha-adrenoceptor characteristics in human and canine prostate. Fed Proc. 1986 Oct;45(11):2609-14. PMID 2428671
- [Background] Hieble JP, Ruffolo RR Jr. The use of alpha-adrenoceptor antagonists in the pharmacological management of benign prostatic hypertrophy: an overview. Pharmacol Res. 1996 Mar;33(3):145-60. doi: 10.1006/phrs.1996.0022. PMID 8880886
- [Background] Madersbacher S, Alivizatos G, Nordling J, Sanz CR, Emberton M, de la Rosette JJ. EAU 2004 guidelines on assessment, therapy and follow-up of men with lower urinary tract symptoms suggestive of benign prostatic obstruction (BPH guidelines). Eur Urol. 2004 Nov;46(5):547-54. doi: 10.1016/j.eururo.2004.07.016. PMID 15474261
- [Background] Wilt TJ, Ishani A, Rutks I, MacDonald R. Phytotherapy for benign prostatic hyperplasia. Public Health Nutr. 2000 Dec;3(4A):459-72. doi: 10.1017/s1368980000000549. PMID 11276294
- [Background] Wilt TJ, Ishani A, Stark G, MacDonald R, Lau J, Mulrow C. Saw palmetto extracts for treatment of benign prostatic hyperplasia: a systematic review. JAMA. 1998 Nov 11;280(18):1604-9. doi: 10.1001/jama.280.18.1604. PMID 9820264
- [Background] Zhu YS, Imperato-McGinley JL. 5alpha-reductase isozymes and androgen actions in the prostate. Ann N Y Acad Sci. 2009 Feb;1155:43-56. doi: 10.1111/j.1749-6632.2009.04115.x. PMID 19250191
- [Background] Crawford ED, Wilson SS, McConnell JD, Slawin KM, Lieber MC, Smith JA, Meehan AG, Bautista OM, Noble WR, Kusek JW, Nyberg LM, Roehrborn CG; MTOPS RESEARCH Group. Baseline factors as predictors of clinical progression of benign prostatic hyperplasia in men treated with placebo. J Urol. 2006 Apr;175(4):1422-6; discussion 1426-7. doi: 10.1016/S0022-5347(05)00708-1. PMID 16516013
- [Background] Boyle P, Gould AL, Roehrborn CG. Prostate volume predicts outcome of treatment of benign prostatic hyperplasia with finasteride: meta-analysis of randomized clinical trials. Urology. 1996 Sep;48(3):398-405. doi: 10.1016/s0090-4295(96)00353-6. PMID 8804493
- [Background] Desgrandchamps F. [Combination therapy in benign prostatic hyperplasia (BPH)]. Ann Urol (Paris). 2004 Dec;38 Suppl 2:S24-8. doi: 10.1016/s0003-4401(04)80003-2. French. PMID 15651487
- [Background] Jacobsen SJ, Jacobson DJ, Girman CJ, Roberts RO, Rhodes T, Guess HA, Lieber MM. Treatment for benign prostatic hyperplasia among community dwelling men: the Olmsted County study of urinary symptoms and health status. J Urol. 1999 Oct;162(4):1301-6. PMID 10492184
- [Derived] Robert G, Descazeaud A, Karsenty G, Saussine C, Azzouzi AR, de la Taille A, Desgrandchamps F, Faix A, Fourmarier M, Georget A, Benard A, Barry Delongchamps N. Prostatic injection of botulinum toxin is not inferior to optimized medical therapy in the management of lower urinary tract symptoms due to benign prostatic hyperplasia: results of a randomized clinical trial. World J Urol. 2018 Jun;36(6):921-929. doi: 10.1007/s00345-018-2193-y. Epub 2018 Jan 30. PMID 29383480